CLINICAL TRIAL: NCT04287868
Title: Phase I/II Trial of Combination Immunotherapy in Subjects With Advanced HPV Associated Malignancies
Brief Title: Combination Immunotherapy in Subjects With Advanced HPV Associated Malignancies
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Charalampos Floudas, MD, DMSc, MS, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 200045; 20-C-0045
Record Dates: First submitted 2020-02-26; First posted 2020-02-27 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-03

CONDITIONS: Cervical Cancer; HPV Cancers; Anal Cancer; Oropharyngeal Cancer; Vulvar, Vaginal, Penile, Rectal Cancer
Keywords: HPV Cancers; HPV Associated Malignancies; Vaccine; Immunotherapy; Immuno-oncology
MeSH Terms: conditions — Uterine Cervical Neoplasms; Anus Neoplasms; Oropharyngeal Neoplasms; Rectal Neoplasms | interventions — NHS-IL12 immunocytokine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1, Arm 1: Human Papillomavirus (HPV) Associated Malignancies (Experimental): Triple Therapy: PDS0101 + NHS-IL12 + M7824 (MSB0011395C); The dose level of NHS-IL12 may decrease depending on dose limiting toxicity (DLT) events. The dose level of human papillomavirus vaccine (HPV) vaccine and M7824 will remain constant.
  If more than 3 of 8 participants have an objective response then accrual will be expanded to 20 evaluable participants.
  Interventions: Biological: PDS0101; Biological: M7824; Biological: NHS-IL12
- Cohort 2, Arm 2: Cervical Cancer With Prior Pelvic Radiation and Boost Brachytherapy (Experimental): Triple Therapy: PDS0101 + NHS-IL12 + M7824 (MSB0011395C); PDS0101 + NHS-IL12 + M7824; Reduced doses.
  May enroll up to 12 participants for a safety evaluation and up to 12 additional participants for preliminary evaluation of efficacy and further evaluation of safety.
  Interventions: Biological: PDS0101; Biological: M7824; Biological: NHS-IL12

INTERVENTIONS:
Biological: PDS0101 — PDS0101 will be administered on Day (D)1, D15, D29 followed by booster vaccines every 4 weeks for up to a year. Subcutaneous 1.0mL (2.4mg of total peptide and 3 mg of R-DOTAP) injection.
Biological: M7824 — M7824 will be administered at a flat dose of 1,200 mg intravenous (IV) (over 1 hour) once every 2 weeks.
  Other Names: MSB0011395C
Biological: NHS-IL12 — NHS-IL12 will be administered at as dose of potentially de-escalating doses by subcutaneous (SC) injection every 4 weeks.

SUMMARY:
Background:

More than 30,000 cases of human papillomavirus (HPV) associated cancers occur annually in the United States. When these cancers spread, they do not respond well to standard treatments and are often incurable. Researchers want to see if a mix of drugs can help.

Objective:

To learn if a mix of immunotherapy drugs can shrink tumors in people with HPV associated cancers.

Eligibility:

People ages 18 and older with locally advanced or metastatic HPV associated cancer, such as cervical cancers; cyclin-dependent kinase inhibitor 2A (P16+) oropharyngeal cancers; anal cancers; vulvar, vaginal, penile, and squamous cell rectal cancers; or other locally advanced or metastatic solid tumors (e.g., lung, esophagus) that are known HPV+ cancers

Design:

Participants will be screened with:

* medical history
* disease confirmation (or tumor biopsy)
* physical exam
* body scans (computed tomography (CT), magnetic resonance imaging (MRI), and/or nuclear)
* blood tests
* electrocardiogram (to measure the electrical activity of the heart)
* urine tests.

Participants will get PDS0101 injected under the skin every 4 weeks for 6 doses. Then they will get it every 3 months for 2 doses.

Participants will get M7824 (MSB0011395C) by intravenous infusion every 2 weeks. For this, a needle is inserted into a vein. The drug is given over a 1-hour period.

Participants will get NHS-IL12 injected under the skin every 4 weeks.

Participants will get the study drugs for up to 1 year. They will visit the NIH every 2 weeks. They will repeat the screening tests during the study.

About 28 days after treatment ends, participants will have a follow-up visit or telephone call. Then they will be contacted every 3 months for 1 year, and then every 6 months after that, for the rest of their life.

Patients with cervical cancer with prior pelvic radiation and boost brachytherapy will be enrolled in a separate cohort to evaluate safety and preliminary evidence of efficacy...

DETAILED DESCRIPTION:
Background:

Metastatic or refractory/recurrent HPV associated malignancies (cervical, anal, oropharyngeal cancers etc.) are poorly palliated by standard therapies. There is an unmet need for active treatments for these tumors.

In a phase I trial of M7824 (MSB0011395C) (NCT02517398) 15 out of 43 (34.9%) participants with HPV associated malignancies had radiographic tumor responses according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 or Immune Response Evaluation Criteria in Solid Tumors (iRECIST).

While the response rate observed with M7824 appears to be higher than single agent programmed cell death protein 1 (PD-1) inhibitors alone (15-20%), the majority of patients with these diseases still do not seem to benefit from immunotherapy.

Preclinical studies suggest that the use of a combination of multiple immunotherapy agents may have improved anti-tumor efficacy.

Specifically, preclinical studies have shown that the combination of three immunotherapy agents (1) a therapeutic vaccine against human papilloma virus (HPV) positive cancers (PDS0101), (2) a bifunctional fusion protein targeting programmed death-ligand 1 (PD-L1) and transforming growth factor (TGF) beta (M7824), and (3) a tumor targeted immunocytokine (NHS-IL12) produces greater anti-tumor activity than any single or dual combination of these agents.

Objective:

To evaluate the objective response rate (ORR) according to Response Evaluation Criteria (RECIST 1.1) of the combination of (1) a therapeutic vaccine against HPV positive cancers (PDS0101), (2) a tumor targeted immunocytokine (NHS-IL12) and (3) a bifunctional fusion protein targeting PD-L1 and TGF beta (M7824) in subjects with checkpoint naive advanced HPV associated malignancies.

Eligibility:

Age >= 18 years old.

Subjects with cytologically or histologically confirmed locally advanced or metastatic HPV associated malignancies:

Cervical cancers;

P16+ Oropharyngeal cancers;

Anal cancers;

Vulvar, vaginal, penile, and squamous cell rectal cancers;

Other locally advanced or metastatic solid tumors (e.g. lung, esophagus) that are known HPV+.

Prior first line systemic therapy is required unless the participant declines standard treatment after appropriate counseling has been provided.

Subjects must have measurable disease.

Design:

This is a phase I/II trial of combination immunotherapy.

The trial will be conducted using a Simon optimal two-stage design.

Participants will receive HPV vaccine + NHS-IL12 + M7824.

The first six participants will be evaluable for dose limiting toxicities (DLTs) and accrual will only continue to 8 participants who have not been treated with checkpoint inhibitors if less than 2 out of the first 6 participants experience a DLT.

If three or more out of eight participants who have not been treated with checkpoint inhibitors have objective responses accrual will be expanded to enroll 20 evaluable participants.

Patients with cervical cancer with prior pelvic radiation and boost brachytherapy will be enrolled in a separate cohort to evaluate safety and preliminary evidence of efficacy.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects with cytologically or histologically confirmed locally advanced or metastatic human papilloma virus (HPV) associated malignancies:

* Cervical cancers;
* cyclin-dependent kinase inhibitor 2A (P16+) Oropharyngeal cancers;
* Anal cancers;
* Vulvar, vaginal, penile, and squamous cell rectal cancers;
* Other locally advanced or metastatic solid tumors (e.g., lung, esophagus) that are known HPV+.

Subjects must have measurable disease, per response evaluation criteria in solid tumors (RECIST) 1.1.

Subjects must have received one prior line of systemic chemotherapy as well as checkpoint therapy if checkpoint therapy is Food and Drug Administration (FDA) approved for that specific tumor type (e.g., head and neck squamous cell carcinoma (HNSCC) and programmed death-ligand 1 (PDL1+) cervical cancer). Prior checkpoint therapy is not needed where checkpoint therapy has not been FDA approved for that specific tumor type (e.g., anal, vaginal, vulvar, penile, PDL1 negative cervical). Exceptions to the above include participant who are not eligible to receive the above therapies or who decline these standard treatment options after appropriate counseling has been provided.

Age >= 18 years.

Eastern Cooperative Oncology Group (ECOG) performance status <= 2.

Adequate hematologic function at screening, as follows:

* Absolute neutrophil count (ANC) >=1 x 10^9/L;
* Hemoglobin >= 9 g/dL;
* Platelets >=75,000/microliter.

Adequate renal and hepatic function at screening, as follows:

* Serum creatinine <= 1.5 x upper limit of normal (ULN) OR Measured or calculated creatinine clearance >=40 mL/min for participant with creatinine levels > 1.5 X institutional ULN (GFR can also be used in place of creatinine or CrCl);
* Bilirubin <= 1.5 x ULN OR in subjects with Gilbert's syndrome, a total bilirubin <= 3.0 x ULN;
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <= 2.5 x ULN, unless liver metastases are present, then values must be <= 3 x ULN).

The effects of the immunotherapies on the developing human fetus are unknown. For this reason and because immunotherapeutic agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use highly effective contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for two months after study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

Participants serologically positive for human immunodeficiency virus (HIV), hepatitis (Hep) B, Hep C are eligible as long as the viral loads are undetectable by quantitative polymerase chain reaction (PCR). HIV positive participants must have clusters of differentiation 4 (CD4) count >= 200 cells per cubic millimeter at enrollment, be on stable antiretroviral therapy for at least 4 weeks and have no reported opportunistic infections or Castleman's disease within 12 months prior to enrollment.

Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

Participants with prior investigational drug, chemotherapy, immunotherapy or any prior radiotherapy (except for palliative bone directed therapy) within the past 28 days prior to the first drug administration except if the investigator has assessed that all residual treatment-related toxicities have resolved or are minimal and feel the participant is otherwise suitable for enrollment. Participants may continue adjuvant hormonal therapy in the setting of a definitively treated cancer (e.g., breast cancer).

Known intolerance to or life-threatening side effects resulting from prior checkpoint inhibitor therapy.

Major surgery within 28 days prior to the first drug administration (minimally invasive procedures such as diagnostic biopsies are permitted).

Known active brain or central nervous system metastasis (less than a month out from definitive radiotherapy or surgery), seizures requiring anticonvulsant treatment (<3 months) or clinically significant cerebrovascular accident (<3 months). In order to be eligible participant must have repeat central nervous system (CNS) imaging at least a month after definitive treatment showing stable CNS disease. Participants with evidence of intra-tumoral or peritumoral hemorrhage on baseline imaging are also excluded unless the hemorrhage is grade <= 1 and has been shown to be stable on two consecutive imaging scans.

Pregnant women are excluded from this study because these drugs have not been tested in pregnant women and there is potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with these immunotherapies, breastfeeding should be discontinued if the mother is treated on this protocol.

Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent with exception of:

* Diabetes type I, eczema, vitiligo, alopecia, psoriasis, hypo- or hyperthyroid disease or other mild autoimmune disorders not requiring immunosuppressive treatment;
* Subjects requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses <= 10 mg of prednisone or equivalent per day;
* Administration of steroids for other conditions through a route known to result in a minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation) is acceptable;
* Subjects on systemic intravenous or oral corticosteroid therapy with the exception of physiologic doses of corticosteroids (<= the equivalent of prednisone 10 mg/day) or other immunosuppressives such as azathioprine or cyclosporin A are excluded on the basis of potential immune suppression. For these subjects these excluded treatments must be discontinued at least 1 weeks prior to enrollment for recent short course use (<= 14 days) or discontinued at least 4 weeks prior to enrollment for long term use (> 14 days). In addition, the use of corticosteroids as premedication for contrast- enhanced studies is allowed prior to enrollment and on study.

Subjects with a history of serious intercurrent chronic or acute illness, such as cardiac or pulmonary disease, hepatic disease, bleeding diathesis or recent (within 3 months) clinically significant bleeding events, or other illness considered by the Investigator as high risk for investigational drug treatment.

Subjects unwilling to accept blood products as medically indicated.

History of non-HPV associated second malignancy within 3 years of enrollment except localized malignancy which has been adequately treated or malignancy which does not require active systemic treatment (e.g., low risk chronic lymphocytic leukemia (CCL). Patients taking adjuvant hormonal therapy for definitively treated cancers (e.g., breast cancer) are eligible.

Subjects with a known severe hypersensitivity reaction to a monoclonal antibodies (grade >/= 3 National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) v5) will be evaluated by the allergy/immunology team prior to enrollment.

Receipt of prior lymphodepleting chemotherapy (e.g., cyclophosphamide, fludarabine) or any organ transplantation requiring ongoing immunosuppression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2026-07-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Charalampos Floudas, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD)recorded in the medical record will be shared with intramural investigators upon request. In addition, all large-scale genomic sequencing data will be shared with subscribers to the database of Genotypes and Phenotypes (dbGaP). All collected IPD will be shared with collaborators under the terms of collaborative agreements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to the Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Genomic data are made available via the database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- [Derived] Floudas CS, Goswami M, Donahue RN, Pastor DM, Redman JM, Brownell I, Turkbey EB, Cordes LM, Steinberg SM, Manu M, Francis DC, Lamping E, Marte JL, Kackley M, Krauss E, Manukyan M, Jochems C, Schlom J, Gulley JL, Strauss J. Novel Combination Immunotherapy and Clinical Activity in Patients With HPV-Associated Cancers: A Nonrandomized Clinical Trial. JAMA Oncol. 2025 Apr 1;11(4):394-399. doi: 10.1001/jamaoncol.2024.6998. PMID 39976981
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-C-0045.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1, Arm 1: Human Papillomavirus (HPV) Associated Malignancies: Cohort 1, Arm 1, Treatment Assignment Code (TAC) 1: Participants with HPV associated malignancies will receive human papillomavirus (HPV) vaccine every (q) 4 weeks x6, then q3 months (MO) x2 + NHS-IL12 q 4 weeks (wks) + M7824 q 2 wks.
  PDS0101 will be administered on Day (D)1, D15, D29 followed by booster vaccines every 4 weeks for up to a year. Subcutaneous 1.0mL (2.4mg of total peptide and 3 mg of R-DOTAP (Versamune) injection).
  M7824 will be administered at a flat dose of 1,200 mg intravenous (IV) (over 1 hour) once every 2 weeks.
  NHS-IL12 will be administered by subcutaneous (SC) injection every 4 weeks.
- Cohort 2, Arm 2: Cervical Cancer With Prior Pelvic Radiation and Boost Brachytherapy: Cohort 2, Arm 2, Treatment Assignment Code (TAC) 1: Participants with cervical cancer with prior pelvic radiation and boost brachytherapy will receive human papillomavirus (HPV) vaccine + NHS-IL12 + M7824 (MSB0011359C) at reduced doses.
  PDS0101 will be administered on Day (D)1, D15, D29 followed by booster vaccines every 4 weeks for up to a year. Subcutaneous 1.0mL (2.4mg of total peptide and 3 mg of R-DOTAP (Versamune) injection).
  M7824 will be administered at a flat dose of 1,200 mg intravenous (IV) (over 1 hour) once every 2 weeks.
  NHS-IL12 will be administered by subcutaneous (SC) injection every 4 weeks.
Period: Overall Study
Arm/Group | Cohort 1, Arm 1: Human Papillomavirus (HPV) Associated Malignancies | Cohort 2, Arm 2: Cervical Cancer With Prior Pelvic Radiation and Boost Brachytherapy
Started | 48 | 3
Completed | 47 | 3
Not Completed | 1 | 0
Not completed — Screening fail | 1 | 0

BASELINE CHARACTERISTICS:
Population: Data was collected and reported here for one participant in cohort 1 who was a screening fail.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1, Arm 1: Human Papillomavirus (HPV) Associated Malignancies | Cohort 2, Arm 2: Cervical Cancer With Prior Pelvic Radiation and Boost Brachytherapy | Total
Number analyzed (Participants) | 48 | 3 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 3 | 40
  >=65 years | 11 | 0 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.54 (10.72) | 51.17 (19.55) | 57.16 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 3 | 24
  Male | 27 | 0 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 0 | 5
  Not Hispanic or Latino | 41 | 2 | 43
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 1 | 7
  White | 37 | 2 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 48 | 3 | 51

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response (BOR) in Checkpoint Naive and Immune Checkpoint Blockade (ICB) Resistant Disease in Participants With Advanced or Metastatic Human Papillomavirus (HPV) Associated Malignancies
Description: BOR is defined as a complete response or partial response assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Complete response is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: Every 2 months, up to approximately 10 months
Population: 48 participants were screened for Cohort (C)1, 1 was a screen fail => 47 were treated on C1. 3 participants were screened for C2 and were treated on it. 50 participants (47 in C1 and 3 in C2) comprise the complete treated population ("All participants"). As pre-specified by the protocol cohort 2 is not required to be reported independently.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: Participants with Human Papillomavirus Associated Malignancies (N = 50, 47 from Cohort 1, 3 from Cohort 2)
- Participants With Human Papillomavirus 16 (HPV16+) Tumors: Participants with Human Papillomavirus 16 Tumors (HPV16+) from both Cohort 1 and Cohort 2 further stratified by prior immune checkpoint blockade.
  (N=37; 34 from Cohort 1, 3 from Cohort 2)
- Human Papillomavirus 16 Tumors (HPV-16+), Immune Checkpoint Blockade (ICB) - Naive: Participants with tumor testing positive for HPV16 and no previous exposure to an immune checkpoint blockade agent.
  (N= 8; 7 from Cohort 1, 1 from Cohort 2)
- Human Papillomavirus 16 Tumors (HPV-16+), Immune Checkpoint Blockade (ICB) - Resistant: Participants with tumor testing positive for HPV16 and disease progression following prior treatment with immune checkpoint blockade agent.
  (N= 29; 27 from Cohort 1, 2 from Cohort 2)
Arm/Group | All Participants | Participants With Human Papillomavirus 16 (HPV16+) Tumors | Human Papillomavirus 16 Tumors (HPV-16+), Immune Checkpoint Blockade (ICB) - Naive | Human Papillomavirus 16 Tumors (HPV-16+), Immune Checkpoint Blockade (ICB) - Resistant
Number analyzed (Participants) | 50 | 37 | 8 | 29
Participants
  Complete Response | 4 | 4 | 2 | 2
  Partial Response | 7 | 7 | 3 | 4
  Overall Response rate (CR+PR) | 11 | 11 | 5 | 6

2. Secondary Outcome: Number of Participants With Grades 1, 2, 3, 4 and/or 5 Treatment Related Adverse Events
Description: Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Grade 1 is mild. Grade 2 is moderate. Grade 3 is severe. Grade 4 is life-threatening. Grade 5 is death related to adverse event.
Time Frame: Date treatment consent signed to date off study, approximately 34 months and 20 days.
Population: Pre-specified in the protocol for cohort 1 only. 1/48 participants in cohort 1 was a screening fail.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Arm 1: Human Papillomavirus (HPV) Associated Malignancies
Number analyzed (Participants) | 47
Participants
  Grade 1 | 45
  Grade 2 | 42
  Grade 3 | 25
  Grade 4 | 1
  Grade 5 | 0

3. Secondary Outcome: Progression-Free Survival (PFS) Time
Description: PFS is defined as the time from the date of first treatment to the date of disease progression or death (any cause) whichever occurs first. Participants who do not have disease progression or have not died at the end of follow up will be censored at the last known date the participant was progression free. Progression was assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Progressive disease is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The appearance of one or more new lesions is also considered progressions.
Time Frame: PFS is defined as the time from the date of first treatment to the date of disease progression or death (any cause) whichever occurs first
Reporting Status: Not Posted, anticipated posting 2026-07

4. Secondary Outcome: Overall Survival (OS)
Description: OS will be evaluated using Kaplan-Meier methods and is defined as the time from the date of first treatment to the date of death (any cause). Participants who are alive at the end of follow up will be censored at the last known date alive.
Time Frame: The time from the date of first treatment to the date of death (any cause)
Reporting Status: Not Posted, anticipated posting 2026-07

5. Secondary Outcome: Ratio of Participants That Are Hospitalized Because of Adverse Events Attributed to Disease Progression.
Description: Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Progressive disease is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The appearance of one or more new lesions is also considered progressions.
Time Frame: While participant on study; an average of 3 months
Measure: Number; unit: Proportion of participants
Arm/Group | Cohort 1, Arm 1: Human Papillomavirus (HPV) Associated Malignancies | Cohort 2, Arm 2: Cervical Cancer With Prior Pelvic Radiation and Boost Brachytherapy
Number analyzed (Participants) | 47 | 3
Proportion of participants | 0.04 | 0

6. Secondary Outcome: Number of Treatment Related Grades 1, 2, 3, 4 and/or 5 Adverse Events
Description: as for outcome 2
Time Frame: Date treatment consent signed to date off study, approximately 34 months and 20 days.
Population: Pre-specified in the protocol for cohort 2 only.
Measure: Number; unit: adverse events
Arm/Group | Cohort 2, Arm 2: Cervical Cancer With Prior Pelvic Radiation and Boost Brachytherapy
Number analyzed (Participants) | 3
adverse events
  Grade 1 | 3
  Grade 2 | 3
  Grade 3 | 1
  Grade 4 | 1
  Grade 5 | 0

7. Secondary Outcome: Duration of Response (DOR)
Description: DOR is measured from the time measurement criteria are met for complete response (CR) or partial response (PR) (whichever is first recorded) until the first date that progressive disease (PD) is objectively documented and is evaluated using the Kaplan-Meier method. Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Complete response is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. Progressive disease is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The appearance of one or more new lesions is also considered progressions.
Time Frame: At disease progression, an average of 10 months
Population: 1/48 participants in cohort 1 was a screening fail.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1, Arm 1: Human Papillomavirus (HPV) Associated Malignancies | Cohort 2, Arm 2: Cervical Cancer With Prior Pelvic Radiation and Boost Brachytherapy
Number analyzed (Participants) | 47 | 3
Months | 10.6 [3.7 to NA] — Not estimable: not enough events to estimate. | 10.2 [NA to NA] — Confidence interval cannot be calculated for one participant.

8. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 34 months and 20 days.
Population: 1/48 participants in cohort 1 was a screening fail.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Arm 1: Human Papillomavirus (HPV) Associated Malignancies | Cohort 2, Arm 2: Cervical Cancer With Prior Pelvic Radiation and Boost Brachytherapy
Number analyzed (Participants) | 47 | 3
Participants | 47 | 3

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 34 months and 20 days.
Description: 1/48 participants in cohort 1 was a screening fail.
Arm/Group | Cohort 1, Arm 1: Human Papillomavirus (HPV) Associated Malignancies | Cohort 2, Arm 2: Cervical Cancer With Prior Pelvic Radiation and Boost Brachytherapy
All-Cause Mortality (participants affected / at risk) | 28/47 | 0/3
Serious Adverse Events (participants affected / at risk) | 18/47 | 1/3
Other Adverse Events (participants affected / at risk) | 47/47 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1, Arm 1: Human Papillomavirus (HPV) Associated Malignancies (N=47) | Cohort 2, Arm 2: Cervical Cancer With Prior Pelvic Radiation and Boost Brachytherapy (N=3)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (4) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (3) | 1 (2)
Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Cardiac disorders - Other, Immune mediated myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Duodenal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 1 (1) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 1 (6) | 0 (0)
General disorders and administration site conditions - Other, Hematuria (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, MUCOSAL BLEEDING, VAGINAL HEMORRHAGE; (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, Mucosal bleeding (General disorders) | 2 (2) | 0 (0)
General disorders and administration site conditions - Other, Mucosal bleeding (anal bleeding) (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, Mucosal bleeding, vaginal (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, Mucosal bleeding-Hematuria (General disorders) | 1 (2) | 0 (0)
Hematuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Immune system disorders - Other, Hemophagocytic Lymphohistiocytosis (Immune system disorders) | 1 (1) | 0 (0)
Infections and infestations - Other, COVID (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1, Arm 1: Human Papillomavirus (HPV) Associated Malignancies (N=47) | Cohort 2, Arm 2: Cervical Cancer With Prior Pelvic Radiation and Boost Brachytherapy (N=3)
Abdominal pain (Gastrointestinal disorders) | 5 (8) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 5 (6) | 0 (0)
Alanine aminotransferase increased (Investigations) | 9 (24) | 1 (3)
Alkaline phosphatase increased (Investigations) | 9 (16) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 31 (126) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 12 (14) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Arterial thromboembolism (Vascular disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (6) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 14 (27) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 3 (3) | 0 (0)
Blurred vision (Eye disorders) | 3 (3) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
CPK increased (Investigations) | 1 (1) | 0 (0)
Cardiac disorders - Other, Immune mediated myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac troponin I increased (Investigations) | 1 (2) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 5 (5) | 0 (0)
Cholesterol high (Investigations) | 3 (3) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 15 (20) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 0 (0)
Creatinine increased (Investigations) | 8 (11) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 9 (10) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 7 (8) | 0 (0)
Dizziness (Nervous system disorders) | 7 (8) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (3) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 0 (0)
Edema face (General disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 4 (6) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 (17) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Eye disorders - Other, (left eye) (Eye disorders) | 1 (1) | 0 (0)
Eye disorders - Other, left eye stye (Eye disorders) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 2 (2) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 2 (3) | 0 (0)
Fatigue (General disorders) | 26 (40) | 1 (3)
Fever (General disorders) | 6 (8) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Flu like symptoms (General disorders) | 30 (65) | 3 (7)
Fracture (Injury, poisoning and procedural complications) | 3 (4) | 0 (0)
GGT increased (Investigations) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, Gastrointestinal disorders - blood in stool (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, blood noted in stool (Gastrointestinal disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, anal hemorrhage (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, (mucosal bleeding): Hematuria (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) — Bleeding from tumor sites: R. armpit and chest (intermittent)
General disorders and administration site conditions - Other, Bleeding gums when brushing teeth (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, Dyschezia (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, Epistaxis (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, Gum Bleeding (General disorders) | 2 (2) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) — Gum bleeding noted in sputum x1 episode
General disorders and administration site conditions - Other, Gum bleeding w/ dental procedure (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, Hematuria (General disorders) | 1 (2) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) — Mocosal bleeding, oral hemorrhage; intermittent bleeding when brushing teeth
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) — Mucosal bleeding,expected; intermittent when brushing teeth
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) — Mucosal bleeding; nasopharynx; intermittent
General disorders and administration site conditions - Other, Mucosal Bleeding - "Bloody BM" (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, Mucosal Bleeding - Gingival (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, Mucosal Bleeding - Hematuria (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, Mucosal Bleeding - TRACH secretions (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) — Mucosal Bleeding -Gingival with brushing teeth
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) — Mucosal Bleeding, Gingival bleed with dental care
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) — Mucosal Bleeding, Intermittent with brushing teeth (Gingival bleed with brushing teeth)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) — Mucosal Bleeding,Transient Hemoptysis in a.m. when awakens
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) — Mucosal Bleeding; Oozing round PEG site
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) — Mucosal Bleeding; Oral hemorrhage; Intermittent gingival bleeding w/ brushing
General disorders and administration site conditions - Other, Mucosal Hemorrhage - Hemoptysis (General disorders) | 1 (2) | 0 (0)
General disorders and administration site conditions - Other, Mucosal bleeding (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, Mucosal bleeding - Epistaxis (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) — Mucosal bleeding,(vaginal bleeding s/sp stent change)
General disorders and administration site conditions - Other, Mucosal bleeding-Hematochezia (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) — Occasional Red spots when wiping after urinating
General disorders and administration site conditions - Other, Rectal Bleeding (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, TRACH secretion (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, Vaginal bleeding (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) — Vaginal hemorrhage; 3 days of vaginal bleeding
General disorders and administration site conditions - Other, anal bleeding (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, bleeding from tumor sites (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) — bleeding from tumor sites: (R. axilla/chest)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) — bleeding vessels on posterior bladder wall
General disorders and administration site conditions - Other, epistaxis (General disorders) | 1 (2) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) — intermittent blood noticed with blowing nose/gum bleeding
General disorders and administration site conditions - Other, intermittent gum bleeding (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, intermittent gum bleeding w/flossing (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, intermittent rectal bleeding (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gum infection (Infections and infestations) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 10 (15) | 0 (0)
Hematuria (Renal and urinary disorders) | 7 (9) | 1 (1)
Hot flashes (Vascular disorders) | 2 (2) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (4) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (5) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 13 (18) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 6 (7) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 3 (10) | 1 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 7 (9) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 7 (8) | 1 (3)
Hypotension (Vascular disorders) | 6 (7) | 1 (1)
Hypothyroidism (Endocrine disorders) | 4 (4) | 0 (0)
Hypoxia (Renal and urinary disorders) | 1 (1) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0)
Infections and infestations - Other, COVID (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, COVID-19 positive (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, Staph Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, at PEG site (Infections and infestations) | 1 (2) | 0 (0)
Infections and infestations - Other, AAA noted on BL CT (Infections and infestations) | 1 (2) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Injection site reaction (General disorders) | 34 (115) | 3 (9)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Investigations - Other, AAA noted on BL CT (Investigations) | 1 (2) | 0 (0)
Investigations - Other, CRP Increased (Investigations) | 2 (2) | 0 (0)
Investigations - Other, Elevated Hgb A1C (Investigations) | 1 (1) | 0 (0)
Investigations - Other, Low iron levels (Investigations) | 1 (1) | 0 (0)
Investigations - Other, Oral lesion (Investigations) | 0 (0) | 1 (1)
Investigations - Other, elevated troponin (Investigations) | 1 (1) | 0 (0)
Laryngeal hemorrhage (Renal and urinary disorders) | 2 (2) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 5 (6) | 0 (0)
Lung infection (Infections and infestations) | 3 (3) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphedema (Vascular disorders) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 21 (48) | 0 (0)
Malaise (General disorders) | 2 (2) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 12 (21) | 0 (0)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, RLE foot drop (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 16 (25) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Benign; Keratoacanthomas, torso
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Keratoacanthoma, Right eyelid; Derm consult to be scheduled at next visit
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Keratoacanthomas - torso, neck, face, scalp
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Polyps (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — torso, front/back, neck. Eruptive Keratoacanthomas
Nervous system disorders - Other, (expressive aphasia) (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorders - Other, Facial tingling (Nervous system disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (2) | 1 (1)
Non cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 7 (7) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Pain (General disorders) | 18 (37) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Paresthesia (Nervous system disorders) | 2 (2) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 1 (2) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 3 (3) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 4 (6) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (4) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (17) | 1 (1)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rash - Eruptive Keratoacanthomas (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 5 (10) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 11 (18) | 0 (0)
Rash pustular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rectal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Renal and urinary disorders - Other, Asymptomatic bacteremia (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal and urinary disorders - Other, urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, SARS-CoV-2 infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Serum amylase increased (Investigations) | 1 (3) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Basal Cell Carcinoma (cheek) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Bruise to R Shin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Dermatitis,bilateral forearms (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Diaphoresis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Diaphoretic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Inguinal pimple (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, KA's back, legs, neck (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Skin and subcutaneous tissue disorders - Other, KA's various parts of the body (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Keratoacanthoma (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Keratoacanthoma nose/hands (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Neck lesion/mass, outside records (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, R elbow/arm rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Seborrheic dermatitis, scalp & beard (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — dermatitis/benign lichenoid keratoses, R hip and L upper back/posterior shoulder
Skin and subcutaneous tissue disorders - Other, itchy blemish on skin of back (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, papule upper, inner right arm (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, rash multiple sites (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin papilloma (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stoma site infection (Infections and infestations) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Superficial thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 2 (2) | 0 (0)
Surgical and medical procedures - Other, (left VATS lower lobe wedge resection x2) (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, (right VATS lower lobectomy) (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, Bifrontal Craniotomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, Cardiac cath (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, Hemorrhoidectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, Upper abdomen midline surgical incision (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, right VATS (Surgical and medical procedures) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (2) | 0 (0)
Testicular disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 3 (3) | 0 (0)
Thrush (Infections and infestations) | 1 (1) | 0 (0)
Thyroid stimulating hormone increased (Endocrine disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (6) | 1 (2)
Urinary tract obstruction (Renal and urinary disorders) | 3 (3) | 0 (0)
Uveitis (Eye disorders) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vascular disorders - Other, Bil PE (Vascular disorders) | 1 (1) | 0 (0)
Vascular disorders - Other, livedo reticularis (Vascular disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 11 (15) | 0 (0)
Weight gain (Investigations) | 1 (2) | 0 (0)
Weight loss (Investigations) | 4 (4) | 0 (0)
White blood cell decreased (Investigations) | 3 (3) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT04287868/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-08): https://cdn.clinicaltrials.gov/large-docs/68/NCT04287868/ICF_001.pdf